CLINICAL TRIAL: NCT01146223
Title: Observational - WT-1's Role in Leukemogenesis
Brief Title: Biomarkers in Bone Marrow Samples From Patients With Acute Promyelocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B7; NCI-2012-02717 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000671471 (Other: Clinical Trials.gov)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Adult Acute Myeloid Leukemia; Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Promyelocytic Leukemia (M3); Childhood Acute Promyelocytic Leukemia (M3)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Basic science (correlative studies): Patient mRNA samples from diagnosis are analyzed via quantitative PCR to measure WT1 and VEGF-1 expression.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is studying biomarkers in patients with acute promyelocytic leukemia. Studying samples of bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and about biomarkers related to cancer.

DETAILED DESCRIPTION:
OBSERVATIONAL STUDY MODEL: Case-only TIME PERSPECTIVE: Retrospective BIOSPECIMEN RETENTION: Samples With DNA BIOSCPECIMEN DESCRIPTION: Bone marrow STUDY POPULATION DESCRIPTION: Primary Care Clinic SAMPLING METHOD: Non-Probability Sample

PRIMARY OBJECTIVES:

I. To measure WT1 and VEGF-1 expression in patients with acute promyelocytic leukemia.

OUTLINE: This is a multicenter study.

Patient mRNA samples from diagnosis are analyzed via quantitative PCR to measure WT1 and VEGF-1 expression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute promyelocytic leukemia [t(15;17) translocation]
* Not specified
* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: acute promyelocytic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
WT1 and VEGF-1 expression | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Moazam, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States